CLINICAL TRIAL: NCT03472196
Title: First in Human Clinical Study to Assess the Safety and Preliminary Performance of NitiNotes' Endoluminal Gastroplasty System (EndoZip) for the Treatment of Obesity
Brief Title: NitiNotes' EndoZip System for the Treatment of Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nitinotes Surgical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CLP-01
Record Dates: First submitted 2018-03-04; First posted 2018-03-21 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2019-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Open label, single arm, open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EndoZip System (Experimental): The Nitinotes EndoZip system is designed to allow for the creation of multiple internal gastric segmentation (4-8) in the stomach by using an endoscopic approach. The system allows the forming of wall-to-wall longitudinal attachments of the anterior and posterior stomach walls, creating multiple strictures within.
  Creation of this segmentation may significantly reduce gastric volume, may affect gastric motility and consequently, reduce weight.
  Interventions: Device: EndoZip System

INTERVENTIONS:
Device: EndoZip System — The Nitinotes EndoZip system is designed to allow for the creation of multiple internal gastric segmentation (4-8) in the stomach by using an endoscopic approach. The system allows the forming of wall-to-wall longitudinal attachments of the anterior and posterior stomach walls, creating multiple strictures within.
  Creation of this segmentation may significantly reduce gastric volume, may affect gastric motility and consequently, reduce weight.

SUMMARY:
This is first-in-man safety and performance feasibility study, aimed to provide initial clinical assessment of safety and effectiveness of the EndoZip in the treatment of obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Subject, male or female, is age 18 to 60 years of age.
2. Subject must be able to understand and be willing to sign an informed consent form.
3. Subject must be willing and able to participate in all aspects of the study and agree to comply with all study requirements for the duration of the study. This includes availability of reliable transportation and sufficient time to attend all follow-up visits.
4. Subject has a BMI of 30-40 kg/m2
5. Have had no significant weight change (±5% of total body weight) during 6 months prior to enrollment
6. Subject must be fully ambulatory, without chronic reliance on walking aids such as crutches, walkers or a wheelchair.
7. Subject must be of sufficient and stable medical and mental health, as evaluated by the Principal Investigator.
8. Subject must have a primary care physician that will manage the subject for any co-morbid conditions throughout the study.
9. Subject must have failed standard obesity therapy of diet, exercise, behavior modification, and pharmacologic agents either alone or in combination.
10. Subject agrees not to have any additional weight loss interventional procedures, such as mammoplasty or abdominal lipoplasty or liposuction, or take any over the counter or prescription weight loss medication for the entire study participation duration
11. Type II Diabetes patients who are treated with oral glucose lowering agent and are stable are acceptable.

Exclusion Criteria:

1. Subject has had previous bariatric, gastric or esophageal surgery; intestinal obstruction; portal gastropathy; gastrointestinal tumors; esophageal or gastric varices, or gastroparesis.
2. Subject has history of/or signs and/or symptoms of gastro-duodenal ulcer disease.
3. Uncontrolled diabetes or change in diabetes medication and/or dosage in the 3 months prior to enrolment
4. Uncontrolled hypertension
5. Subject with heart failure, NYHA grade 2 and above.
6. Subject has pre-existing respiratory disease, such as chronic obstructive pulmonary disease (COPD), pneumonia or cancer.
7. Subject has significant esophageal disease including Zenker's diverticulum, severe gastro-esophageal reflux disease (GERD), stricture, Barrett's esophagus, esophageal cancer, esophageal diverticulum, dysphagia, achalasia, or symptoms of dysmotility, which is not controlled with medication.
8. Subject has renal and/or hepatic insufficiency/disease (creatinine above 1.5 mg/dL)
9. Subject has thyroid disease, which is not controlled with medication.
10. Subject is diagnosed with ostocorticular pain, pre-neoplastic lesions or coagulation conditions that may prevent him/her from undergoing a surgical procedure.
11. Subject has a history of intestinal strictures or adhesions and/or any condition that could preclude passage of endoluminal instruments.
12. Female subject who is pregnant (i.e., has a positive urine or blood pregnancy test prior to device use), is suspected to be pregnant, is lactating or is of childbearing potential but refuses to use adequate contraception during the study.
13. Subject is diagnosed with a coagulation disorder.
14. Subjects undergoing chronic steroid therapy.
15. Subjects undergoing immunosuppressive therapy.
16. Subjects who cannot discontinue either prescription or over the counter weight loss medications for at least 30 days prior to the procedure as well as during the trial period.
17. Subjects who have known hiatal hernias greater than 5 cm.
18. Subjects who have poorly controlled psychiatric disease including but not limited to manic-depressive disorder, schizophrenia, borderline personality disorder, depression or suicidal tendencies.
19. Subject has active Crohn's disease or Colitis.
20. Subject currently uses or has a history of illicit drug(s) or abuses alcohol (defined as regular or daily consumption of more than 4 alcoholic drinks per day).
21. Subject has participated in a clinical study with an investigational new drug, biological, or therapeutic device within 6 months prior to enrollment in this study, and does not agree to abstain from participation in other clinical trials of any kind during this study and their participation may interfere with the current study.
22. Subject has any condition that, at the discretion of the investigator, would preclude participation in the study.
23. Unstable diabetes patients who are treated with insulin.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-05-08 (Actual)

PRIMARY OUTCOMES:
Primary - Serious Adverse Events | 6 months
  Incidence of device related SAEs within 6 months post procedure

SECONDARY OUTCOMES:
Efficacy - Suture Durability | 6 months
  Success rate at 6 months after procedure by assessment of the stitches durability / gastroplasty shape in the stomach, to be determined by the investigator using endoscopy and/or Barium X-ray (per physician discretion) at pre-determined intervals.
Efficacy - % Excess Weight Loss (EWL) | 6 months
  %EWL after 6 months from baseline

OTHER OUTCOMES:
Exploratory - Waist Circumference | 6 months
  Change in waist circumference from baseline to 6 months post procedure.
Exploratory - Quality Of Life Questionnaire | 6 months
  Subject change in Patient Assessment of Upper Gastrointestinal Disorders Quality of Life questionnaire (PAGI-QoL) total score from baseline to 6 months post procedure. Total score ranges from 0 (best score) to 45 (worst score).
Exploratory - % Total Body Weight Loss (TBWL) | 6 months
  %TBWL after 6 months from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario HM Sanchinarro, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopez-Nava G, Asokkumar R, Rull A, Fernandez-Corbelle, Bautista I, Dayyeh BA. Safety and Feasibility of a Novel Endoscopic Suturing Device (EndoZip TM) for Treatment of Obesity: First-in-Human Study. Obes Surg. 2020 May;30(5):1696-1703. doi: 10.1007/s11695-019-04370-w. PMID 31898051